CLINICAL TRIAL: NCT01287546
Title: A Phase 1 Study of LY2875358 in Patients With Advanced Cancer
Brief Title: A Study of LY2875358 in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13298; I4C-MC-JTBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — emibetuzumab; Erlotinib Hydrochloride; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2875358 (Experimental)
  Interventions: Drug: LY2875358
- LY2875358 + erlotinib (Experimental)
  Interventions: Drug: LY2875358 + erlotinib
- LY2875358 at Part A highest dose (Experimental)
  Interventions: Drug: LY2875358 at Part A highest dose
- LY2875358 at Part A highest dose + trametinib (Experimental)
  Interventions: Drug: LY2875358 at Part A highest dose + trametinib

INTERVENTIONS:
Drug: LY2875358 — Part A Dose escalation of LY2875358 administered intravenously (IV), Day 1 and 15 every 28 days for at least two cycles.
  Arms: LY2875358
Drug: LY2875358 + erlotinib — Part A2 Dose escalation of LY2875358 administered IV, on Day 1 and 15 every 28 days for at least two cycles in combination with daily erlotinib dosing (150 mg) taken orally (PO).
  Arms: LY2875358 + erlotinib
Drug: LY2875358 at Part A highest dose — Part B (Dose Exploration): LY2875358 at Part A highest dose administered IV, on Day 1 and 15 every 28 days for at least two cycles.
  Arms: LY2875358 at Part A highest dose
Drug: LY2875358 at Part A highest dose + trametinib — Part B (in combination with trametinib): LY2875358 at Part A highest dose administered IV, on Day 1 and 15 every 28 days for at least two cycles, in combination with trametinib at 2 mg orally once daily
  Arms: LY2875358 at Part A highest dose + trametinib

SUMMARY:
The objective of this study is to determine a recommended Phase 2 dose range of LY2875358 that may be safely administered to participants with advanced cancer. In Part A and Part A2 of this study, escalating doses of LY2875358 as monotherapy and in combination with erlotinib will be evaluated for safety and tolerability, respectively. Part B is a dose-confirmation segment for LY2875358 therapy in 5 different types of cancer: nonsquamous non-small cell lung cancer (NSCLC), castrate resistant prostate cancer (CRPC) with bone metastases, renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), or uveal melanoma with liver metastases, and for LY2875358 in combination with trametinib in participants with uveal melanoma with liver metastases.

DETAILED DESCRIPTION:
Protocol amendment (November, 2013) expanded Part B to study LY2875358 in combination with trametinib in participants with uveal melanoma with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Have histological or cytological evidence of cancer (solid tumor, lymphoma, or multiple myeloma) that is advanced and/or metastatic and an appropriate candidate for experimental therapy
* Part A2: Histologic or cytologic diagnosis of advanced Non Small Cell Lung Cancer (NSCLC), Stage IIIB with malignant pleural effusion or Stage IV, completed at least 1 prior systemic regimen, and eligible for erlotinib therapy.
* Part B: Candidate for experimental therapy after standard therapies used or non-eligible for standard therapies. Histological or cytological evidence of 1 of the 5 tumor types:
* Castrate-resistant prostate cancer (CRPC) with bone metastasis:

  --Progressive Disease in the setting of castrate level of testosterone
* Renal Cell Carcinoma (RCC):

  --Histologic diagnosis of either clear-cell or papillary RCC (metastatic and unresectable, or bilateral, multifocal, unresectable RCC localized to kidneys).
* NSCLC:

  --Histologic or cytologic diagnosis of advanced NSCLC, Stage IIIB with malignant pleural effusion or Stage IV
* Hepatocellular Carcinoma (HCC)

  --Histologic or cytologic diagnosis of hepatocellular carcinoma
* Uveal Melanoma with liver metastasis
* Part A: Have the presence of measurable or nonmeasurable disease as defined by the RECIST v1.1 (Eisenhauer et al. 2009) or Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007) or have measureable disease for multiple myeloma.
* Part A2 & B (RCC, NSCLC, HCC, and uveal melanoma): Have measurable disease as defined by RECIST v1.1.
* Give written informed consent prior to any study-specific procedures.
* Adequate organ function.
* Performance status of less than or equal to 2 on ECOG scale.
* Discontinued all previous cancer therapies, and any agents that have not received regulatory approval, for at least 21 days and recovered from the acute effects of therapy. Must have discontinued mitomycin-C or nitrosourea therapy for at least 42 days.
* Reliable and available for the duration of the study and willing to follow study procedures.
* Males and females (reproductive potential): Use medically approved contraceptive precautions during the study and for 4 months following the last dose of study drug.
* Females (childbearing potential): Have had a negative serum pregnancy test before the first dose of study drug and not be breast-feeding.
* Estimated life expectancy that will permit the participants to complete 8 weeks of treatment.

Exclusion Criteria:

* Serious preexisting medical conditions
* Symptomatic central nervous system malignancy or metastasis (screening not required).
* Acute or chronic leukemia.
* Active infection including HIV, hepatitis A, B or C
* Have second primary malignancy that may affect the interpretation of results.
* Have received a liver transplant, or have liver cirrhosis with a Child-Pugh Stage of B or C.
* Patients with active alcohol abuse, as determined by the treating investigator.
* Part A2: Unable to swallow tablets. Intolerant of therapy with erlotinib. Concomitant treatment with the cytochrome P450 3A (CYP3A) modulators. Must not have received treatment with any of these modulators within 14 days of study treatment.
* Have a history of New York Heart Association class ≥3, unstable angina, myocardial infarction 6 months prior to study drug
* QTc greater than 470 msec.
* Received previous treatment with any c-MET experimental therapeutic.
* Part B Expansion Cohort 1 (CRPC):

  1. Increasing use of daily doses of opioid analgesics within 28 days prior to enrollment in the study.
  2. Neuroendocrine prostate cancer.
  3. Patients who have a solitary bone metastasis that has been irradiated are not eligible.
* Part B Expansion Cohort 6 (LY2875358 plus trametinib in participants with uveal melanoma with liver metastasis): Contra-indications for trametinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2010-04-13 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 dose range of LY2875358 monotherapy and in combination with erlotinib | Baseline through Cycle 1

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration (Cmax) | Days 1, 2, 4, 5, 6, 8, 15, and 22 of Cycle 1. Days 1, 15, and 22 of Cycle 2. Days 1 and 15 of Cycles 3 and beyond, as well as 14 days, 29 days, and 57 days following the final treatment
Number of participants with a tumor response | Baseline to study completion (12 months)
Pharmacokinetics: Area under the concentration-time curve (AUC) | Days 1, 2, 4, 5, 6, 8, 15, and 22 of Cycle 1. Days 1, 15, and 22 of Cycle 2. Days 1 and 15 of Cycles 3 and beyond, as well as 14 days, 29 days, and 57 days following the final treatment
Time to progression and overall survival | Baseline to study completion (12 months)
Pharmacokinetics: Area under the concentration-time curve (AUC) of erlotinib or trametinib in combination with LY2875358 | Cycle 1
Change from baseline in Brief Pain Inventory (BPI) in Part B: Expansion Cohort 1 | Baseline to study completion (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - University of California - San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Univ of California San Francisco, San Francisco, California
  - UCLA, Santa Monica, California
  - Mayo Clinic of Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson University, Philadelphia, Pennsylvania